CLINICAL TRIAL: NCT00226369
Title: Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy/Safety of CY-1503 (Cylexin) in Prevention of Reperfusion Injury in Neonates/Infants Undergoing Hypothermic Cardiopulmonary Bypass
Brief Title: Cylexin for Reduction of Reperfusion Injury in Infant Heart Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: X04-01-007R
Record Dates: First submitted 2005-09-21; First posted 2005-09-27 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2005-09

CONDITIONS: Congenital Heart Defects
Keywords: Pediatric; Cardiopulmonary bypass; Congenital heart disease; Reperfusion injury
MeSH Terms: conditions — Heart Defects, Congenital; Reperfusion Injury | interventions — CY 1503

INTERVENTIONS:
Drug: CY-1503

SUMMARY:
We conducted a multicenter, randomized, placebo-controlled trial of Cylexin, an inhibitor of the attachment of white blood cells to the endothelium. Our study population was neonates and infants undergoing hypothermic cardiopulmonary bypass during surgical repair or palliation of congenital heart defects.

DETAILED DESCRIPTION:
Ischemia/reperfusion (I/R) injury is an important adverse effect of cardiopulmonary bypass (CPB) in infants undergoing cardiac surgery. We performed a multicenter, randomized, placebo-controlled, double-blinded trial of the leukocyte-endothelial cell adhesion inhibitor Cylexin in young infants to determine if it reduces I/R injury following hypothermic CPB. Entry criteria included age at surgery 1-45 days, birth weight > 2.3 kg, and planned repair or palliation of congenital heart defects with CPB. We excluded patients with specified antecedent events or conditions, including lung or kidney disease, seizures, necrotizing enterocolitis, infection, or other serious noncardiac morbidity. Randomization was stratified by study center and cardiac diagnosis. Cylexin was administered continuously from sternotomy until 24 hours post CPB. Centers followed their usual operative and postoperative care practices. From December 1997-March 1999, we enrolled 230 infants, 155 for 2-ventricle repairs (Group 1: D-TGA=90, VSD=16, TOF/truncus=22, TAPVR=9, VSD with aortic arch obstruction=18) and 75 for stage 1 palliation (Group 2: single ventricle with aortic arch obstruction). Of those enrolled, 117 were assigned to Cylexin (Group 1=80, Group 2=47) and 113 to placebo (Group 1=75, Group 2=38). Pre- and intraoperative variables were comparable between treatment groups. Early (30 day) mortality for Cylexin versus placebo patients in Group 1 was 0% versus 3.8% (p=0.25) and for Group 2 was 10.8% versus 28.9% (p=0.08). In both risk groups, treatment with Cylexin did not significantly improve other early postoperative outcomes or decrease the occurrence of adverse events. Cylexin did not significantly improve early mortality or postoperative recovery in Group 1 patients. Despite a small sample size, early mortality in Group 2 Cylexin-treated patients tended to be lower, suggesting the need for future trials of agents that could reduce I/R injury in high-risk infants.

ELIGIBILITY:
Inclusion Criteria:1) scheduled cardiac surgery with hypothermic CPB to repair either D-transposition of the great arteries (D-TGA) with intact ventricular septum (IVS) or ventricular septal defect (VSD), VSD with or without aortic arch obstruction (AAO), tetralogy of Fallot (TOF) with or without pulmonary atresia (PA), truncus arteriosus, total anomalous pulmonary venous return (TAPVR), or double outlet right ventricle (DORV), or to palliate hypoplastic left heart syndrome (HLHS) or other forms of single ventricle (SV) with AAO using the stage I (Norwood) operation, 2) age 1-45 days at surgery, 3) birth weight > 2.3 kg, and 4) a cranial ultrasound < 1 week prior to enrollment showing at most grade II hemorrhage in high risk patients -

Exclusion Criteria:Exclusion criteria included the following: 1) need for urgent cardiac surgery, 2) cardiac arrest ≤ 1 week before surgery, 3) prior procedure with hypothermic CPB, 4) acute or chronic infection, 5) major noncardiac congenital anomalies or chromosomal abnormalities, 6) preoperative arterial pH ≤ 7.0, 7) any significant noncardiac organ dysfunction such as renal failure, respiratory failure, seizures, or necrotizing enterocolitis, and 8) use of another investigational drug.

-

Max Age: 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 242
Dates: Start 1997-12; Study Completion 2001-06

PRIMARY OUTCOMES:
1) non-operative mortality within 30 days, 2) time from ICU admission to extubation, 3) 48-hour Ccr, 4) time to eligibility for ICU discharge, and 5) total inotrope score

SECONDARY OUTCOMES:
1) A-a O2 gradient during the first 48 hours 2) total urine output in the first 72 hours, 3) total fluid balance during the first 72 hours, and 4) time to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jane W Newburger, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States